CLINICAL TRIAL: NCT05786092
Title: The Role of Home Telemonitoring in the Evaluation of Patients With Severe Obesity After a Period of Residential Metabolic Rehabilitation.
Brief Title: Impact of Telemonitoring on Metabolic Variables in Severe Obesity
Acronym: teleob
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18C020
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Severe Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment (Experimental)
  Interventions: Device: Telemonitoring
- control (No Intervention)

INTERVENTIONS:
Device: Telemonitoring — Monitoring of the required parameters by means of the data provided by the devices used by patients. The data (weight, body composition, blood pressure, oxygen saturation, physical activity, heart rate and blood glucose) collected according to the predetermined schedule are then saved in a cloud accessible to researchers.
  Arms: treatment

SUMMARY:
The goal of this clinical trial is to compare, in a population of severely obese patients, two different kinds of follow-up after discharge from in-hospital rehabilitation programme.

The main questions addressed are:

* primary outcome: comparing the dropout rate at month 11 of patients followed-up by a telemedicine methodology with that of a traditional outpatient visit follow-up.
* secondary outcome: comparing the amount of weight loss at month 11 in patients followed-up by telemedicine with that registered in patients followed-up by traditional outpatient visits.

Participants are given a set of instruments (scale, activity tracker, automatic blood pressure monitor, oxymeter, and glucometer) and asked to measure vital parameters following a predetermined schedule for one year. Subjects are asked to engage in regular physical activity and follow the nutritional guidelines received at the moment of discharge from hospital.

ELIGIBILITY:
Inclusion Criteria:

* BMI 38-60 kg/m2,
* age between 18 and 65 years,
* patient residing in Piedmont, Lombardy
* Recent admission to San Giuseppe Hospital in Piancavallo for a period of residential rehabilitation.
* Patient with wi-fi and/or mobile data connection at home.

Exclusion Criteria:

* illiteracy
* inability to engage in physical activity
* psychiatric illnesses capable of impairing the proper use of the devices provided by telemonitoring
* cognitive impairment, mental retardation
* predictability of long periods of stay abroad
* anticipation or planning of pregnancy during the year following discharge
* legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
+ dropout rate at month 11 of patients followed-up by a telemedicine methodology with that of a traditional outpatient visit follow-up. | 12 months
  Percentage of patients still in care at month 11 after discharge in each of the two subgroups.

SECONDARY OUTCOMES:
amount of weight loss at month 11 in patients followed-up by telemedicine with that registered in patients followed-up by traditional outpatient visits. | 12 months
  Percentage of patients with weight loss of at least 5% and percentage of patients with weight loss between 0% and 5% at month 11 in each of the two subgroups.

OTHER OUTCOMES:
changes in blood pressure registered at month 11 in patients followed-up by telemedicine and in patients undergoing traditional outpatient visit follow-up. | 12 months
  Variation in blood pressure between the time of discharge and 11 months in patients undergoing the two different strategies in studies
changes in heart rate registered at month 11 in patients followed-up by telemedicine and in patients undergoing traditional outpatient visit follow-up. | 12 months
  Variation in heart rate between the time of discharge and 11 months in patients undergoing the two different strategies in studies
changes in oxygen saturation registered at month 11 in patients followed-up by telemedicine and in patients undergoing traditional outpatient visit follow-up. | 12 months
  Variation in oxygen saturation between the time of discharge and 11 months in patients undergoing the two different strategies in studies
changes in blood glucose registered at month 11 in patients followed-up by telemedicine and in patients undergoing traditional outpatient visit follow-up. | 12 months
  Variation in blood glucose between the time of discharge and 11 months in patients undergoing the two different strategies in studies

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Oggebbio, VCO, Italy